CLINICAL TRIAL: NCT00349089
Title: Adjuvant Chemotherapy With Pemetrexed and Cisplatin vs. Vinorelbine and Cisplatin in NSCLC IB, IIA, IIB, T3N1: a Randomized Phase II Study
Brief Title: Trial on Refinement of Early Stage Lung Cancer Adjuvant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thoraxklinik-Heidelberg gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREAT; 2005-004840-30 (EudraCT Number)
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; adjuvant therapy; clinical feasibility rate
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cisplatin/Vinorelbine
  Interventions: Drug: Cisplatin; Drug: Vinorelbine
- 2 (Experimental): Cisplatin/Pemetrexed
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 d1 and Cisplatin 75 mg/m2 d1; q d22
  Arms: 2
Drug: Cisplatin — Pemetrexed 500 mg/m2 d1 and Cisplatin 75 mg/m2 d1; q d22
  Comparator:
  Vinorelbine 25 mg/m2 d1, 8, 15, 22; q d29 Cisplatin 50 mg/m2 d1, 8; q d29
Drug: Vinorelbine — Vinorelbine 25 mg/m2 d1, 8, 15, 22; q d29
  Arms: 1

SUMMARY:
The purpose of this randomized phase II trial is to determine the clinical feasibility - in terms of patients without dose limiting toxicities or premature treatment withdrawal or death - of the combination of Cisplatin and Pemetrexed and of the combination of Cisplatin and Vinorelbine. The combination of Cisplatin / Pemetrexed is assumed to be distinctly less toxic than Vinorelbine / Cisplatin.

DETAILED DESCRIPTION:
Derived from recent large randomized clinical trials, there is clear evidence for adjuvant chemotherapy in stage IB-IIB (incidental IIIA) non-small cell lung cancer (Arriagada et al., 2004; Winton et al., 2005, Strauss et al., 2004, Douillard et al., 2005). The majority of patients in the adjuvant treatment setting received a combination of Cisplatin and Vinorelbine (Aragiada et al., 2004; Winton et al., 2005; Douillard et al., 2005). This combination improved 5 year-survival rates up to 15% (54% to 69%) (Winton et al., 2005). However, the combination of Cisplatin and Vinorelbine resulted in rates of grade 3/4 neutropenia of around 75%, rates of febrile neutropenia of up to 12.5% and rates of treatment related death of 1-2%. Up to 77% of the patients had at least one dose reduction or omission and 55% required one dose delay or more, most related to neutropenia. Only about 50 % of patients randomized on the combination of cisplatin and vinorelbine received the intended dose of Vinorelbine (dose reduction mainly due to toxicity) and only 50% of patients completed all four cycles of chemotherapy (Winton et al., 2005, Douillard et al., 2005, Alam et al., 2005).

Therefore it seems reasonable to test a less toxic regimen also in early stages after R0 resection of the tumor, where reduced toxicities might improve the feasibility of drug delivery, compliance and the convenience of treatment for the patient and hence perhaps survival.

Pemetrexed, a folate antimetabolite, shows clear activity in non-small cell lung cancer with several Phase II studies of Pemetrexed in combination with Cisplatin, Oxaliplatin, or Carboplatin showing efficacy similar to other standard platinum doublets, with response rates of 27% to 45% and median survival of 8.9 to 10.9 months (Scagliotti et al., 2005; Clarke et al., 2002; Rusthoven et al., 1999; Manegold et al., 2000; Shepherd et al., 2001). The combination of platin and Pemetrexed can be easily delivered and is well tolerated. Furthermore, it only results in a 25% rate of grade 3/4 neutropenia and in vitamin supplemented patients the incidence of febrile neutropenia was < 1%. Dose reductions occur only in 2-4% of the patients and dose delivery of the intended Pemetrexed and platin dose is excellent with dose deliveries of Pemetrexed up to 95% (Hanna et al., 2004; Vogelzang et al., 2003, Scagliotti et al., 2005).

In this randomized phase II trial, the clinical feasibility of the combination of Cisplatin and Pemetrexed as well as of the combination of Cisplatin and Vinorelbine will be assessed. Treatment is considered to have clinical feasibility if dose limiting toxicity will not be observed, and no non-acceptance by the patient leading to premature withdrawal, and no death due to cancer or cancer therapy will occur.

Patients will be randomized according to center, lobectomy vs. pneumonectomy and N0 vs. N1 to 4 cycles (arm A) of 500 mg/m2 pemetrexed d1, and Cisplatin 75 mg/m2 d1, q d22 versus (arm B) 25 mg/m2 Vinorelbine d1, 8, 15, 22, and Cisplatin 50 mg/m2 d1+8; q d29. Radiotherapy or maintenance therapy are not intended. Study drug administration will begin on d28 to d42 after R0 resection of the tumor and within 14 days after randomization.

In an initial study phase 36 patients (i.e. 18 in each treatment arm) will be accrued to confirm feasibility. In the second step, further patients will be recruited up to a total number of 134 (i.e. 67 cases per treatment arm). Patients will be followed-up in 3 monthly intervals for the first 2 years starting 30 days after end of the last cycle and in the 3rd year patients will be followed-up in 6 monthly intervals.

ELIGIBILITY:
Inclusion criteria:

* Histopathologically confirmed diagnosis of non-small cell lung cancer (NSCLC), pathologic stage IB, IIA, IIB or T3N1 (without need for further radiotherapy).
* Complete tumor resection without detectable residual tumor including negative margins (R0) and systematic intraoperative dissection of mediastinal lymph nodes of course lymph node dissection has to comprise all lymph node levels to be removed with standard right or left sided resection. The dissection has to assure the removal of mediastinal lymph nodes more than 1,5 cm on the preoperative CT scan.
* Study drug administration should only be administered to patients with full recovery after surgery and is to begin on d28 to d42 postoperatively
* The following histological tumor types are eligible:
* Squamous Cell Carcinoma
* Adenocarcinoma (including adenocarcinomas with bronchioloalveolar differentiation)
* Large Cell Carcinoma (excluding tumors with slight areas of small cell carcinoma)
* Mixed Cell Carcinoma without small cell fraction
* Provision of informed consent according to local regulatory requirements for participation in the study
* Age ≥ 18 years; < 75 Years
* Karnofsky Performance Status 80% or ECOG 1
* Adequate hematological laboratory parameters
* Hemoglobin 10 g/dl
* ANC 1500/µl
* Platelets 100000/µl
* Adequate hepatic laboratory parameters
* Bilirubin 1.5 x UNL (UNL=Upper Normal Limit )
* ASAT/ALAT 2 x UNL
* Adequate renal laboratory parameters
* Creatinine 1,5 mg/dl and
* Calculated Creatinine Clearance 60 ml/min
* Cardiac function allowing cisplatin chemotherapy (in case of doubt echocardiography is mandatory documenting LVEF >49%)
* Electrocardiogram without significant cardiac arrhythmia
* FEV1 1.2 l post-operatively
* Respiratory function not impeding Cisplatin-based chemotherapy assessed by either absolute DLCO or capillary / arterial BGA in resting condition (absolute DLCO > 40 % or pO2 >60 mmHg in resting condition)
* Agreement by the patient to use an effective method of contraception
* Negative pregnancy test for women of childbearing potential unless they are postmenopausal at baseline. (Postmenopausal women must have been amenorrheic at least for 12 months to be considered of non childbearing potential)

Exclusion criteria:

* Presence of a Pancoast tumor
* Involvement of N2/N3 lymph nodes
* Distant metastases
* The following histological tumor types are excluded
* Pure bronchioloalveolar carcinoma
* Mixed cell carcinoma with small cell fractions
* Large Cell Carcinoma with areas of small cell carcinoma
* Pregnancy or lactation period
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of a CIS of the cervix or non-melanomatous skin cancer. Patients curatively treated and free of disease for at least 5 years will be discussed with the Principal Investigator (LKP) before inclusion.
* Radio- and/or chemotherapy within the last five years
* Concurrent administration of any other antitumor therapy
* Patients who are not compliant with vitamin (folic acid and vitamin B12) intake or to whom administration is not possible
* Hypersensitivity to Pemetrexed or to any of the excipients of Alimta®
* Hypersensitivity to Cisplatin or to any other platinum compound
* Hypersensitivity to Vinorelbin or to any other vinca-alkaloid
* Patient has previously completed or withdrawn from this study or any other study with the respective medication in this study
* Treatment with an investigational new drug, currently or within the last 30 days, and/or participation in another clinical trial, currently or during the last 12 weeks, and/or previous participation in this study
* History of a psychological illness or condition such as to interfere with the patient s ability to understand the requirements of the study
* Patients with any clinically significant disease that in the opinion of the investigator is likely to put the patient at risk or to interfere with the evaluation of the patient's safety and of the study outcome. This includes, but is not limited to:
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 6 months
* Uncontrolled hypertension
* Interstitial pneumonia or extensive or symptomatic interstitial fibrosis of the lung
* pleural effusion or ascites, which cause respiratory compromise. Patients with sero(pneumo)-thorax after hemi-pneumonectomy or lobectomy will not be excluded. Those patients must be monitored for toxicity closely
* Any other active or uncontrolled infection
* Organ allografts
* Patients with neurologic disorders
* A history or presence of any CNS disorder or psychiatric disability judged by the Investigator to be clinically significant and/or interfering with compliance
* A serious concomitant systemic disorder (e.g. active infection including HIV) that in the opinion of the investigator would compromise the patient s ability to complete the study
* Post-operative complications or other surgery-related conditions that could interfere with a study participation
* Hearing function / tinnitus impeding chemotherapy with Cisplatin and / or Vinorelbine
* Alcohol and/or drug abuse
* Patient is unable to interrupt high dose salicylates (like aspirin) or other non-steroidal anti-inflammatory drugs (NSAID´s) for a 5-day period starting 2 days before administration of Pemetrexed (8-day period for long-acting agents such as piroxicam)
* Patients who cannot be regularly observed for psychological, sociological or geographical reasons or other concomitant conditions not permitting adequate follow-up and compliance to the protocol

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-04-14 (Actual)

PRIMARY OUTCOMES:
To determine the clinical feasibility rate of 4 cycles of adjuvant chemotherapy with Pemetrexed and Cisplatin vs. Vinorelbine and Cisplatin | 4 month

SECONDARY OUTCOMES:
To determine and compare the drug delivery between both treatment arms | 4 month
To determine the Time to Treatment Failure (TTTF) | 3 years
To determine the Distant Metastases Free Survival (DMFS) | 3 years
To determine the Local Relapse Free Survival (LRFS) | 3 years
To determine the Overall Survival (OS) | 3 years
To determine the Localization of Relapse | 3 years
To determine dose delivery | 3 years
To determine the Relapse Free Survival (RFS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thomas, Prof. Dr., Principal Investigator — Clinic for thoracic diseases at the University of Heidelberg, Germany; Michael Kreuter, Dr., Study Chair — Clinic for thoracic diseases at the University of Heidelberg, Germany; Johan Vansteenkiste, Prof. Dr., Study Chair — Department of Pulmonology (Respiratory Tumor Unit), University Hospital Gasthuisberg, Catholic University Leuven, Belgium; Frank Griesinger, Prof. Dr., Study Chair — Department of Hematology and Oncology, Oldenburg, Germany.
Locations (14):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Department of Pulmonology (Respiratory Tumor Unit), University Hospital Gasthuisberg, Catholic University Leuven, Belgium., Leuven
- Germany (11):
  - Helios-Klinikum Emil von Behring, Berlin
  - Klinikum Bremen-Ost, Bremen
  - Westdeutsches Tumorzentrum, Essen
  - Department of Hematology and Oncology, University of Göttingen, Göttingen
  - Lungenzentrum Großhansdorf, Großhansdorf
  - Clinic for thoracic diseases at the University of Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Klinik Löwenstein, Löwenstein
  - University of München, München
  - Oldenburg Hospital, Oldenburg
  - Dr. Horst Schmidt Klinik, Wiesbaden
- Centre Hospitalier du Luxembourg, Luxembourg, Luxembourg

REFERENCES:
- [Background] Winton T, Livingston R, Johnson D, Rigas J, Johnston M, Butts C, Cormier Y, Goss G, Inculet R, Vallieres E, Fry W, Bethune D, Ayoub J, Ding K, Seymour L, Graham B, Tsao MS, Gandara D, Kesler K, Demmy T, Shepherd F; National Cancer Institute of Canada Clinical Trials Group; National Cancer Institute of the United States Intergroup JBR.10 Trial Investigators. Vinorelbine plus cisplatin vs. observation in resected non-small-cell lung cancer. N Engl J Med. 2005 Jun 23;352(25):2589-97. doi: 10.1056/NEJMoa043623. PMID 15972865
- [Background] Alam N, Shepherd FA, Winton T, Graham B, Johnson D, Livingston R, Rigas J, Whitehead M, Ding K, Seymour L. Compliance with post-operative adjuvant chemotherapy in non-small cell lung cancer. An analysis of National Cancer Institute of Canada and intergroup trial JBR.10 and a review of the literature. Lung Cancer. 2005 Mar;47(3):385-94. doi: 10.1016/j.lungcan.2004.08.016. PMID 15713522
- [Background] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Background] Strauss G, Herndon J, Maddaus MA, et al. Randomized clinical trial of adjuvant chemotherapy with Paclitaxel and Carboplatin following resection in stage I B non-small cell lung cancer (NSCLC): Report of Cancer and Leukaemia Group B (CALGB) protocol 9633. Proc Am Soc Clin Oncol 22: 621 (# 7019)2004
- [Background] Douillard J, Rosell R, Delena M, et al. ANITA: Phase III adjuvant Vinorelbine and Cisplatin versus observation in completely resected (stage I-III) non-small lung cancer patients: Final results after 70-month median follow up. Proc Am Soc Clin Oncol 23: 624 (# 7013) 2005
- [Derived] Kreuter M, Vansteenkiste J, Griesinger F, Hoffmann H, Dienemann H, De Leyn P, Thomas M. Trial on refinement of early stage non-small cell lung cancer. Adjuvant chemotherapy with pemetrexed and cisplatin versus vinorelbine and cisplatin: the TREAT protocol. BMC Cancer. 2007 May 8;7:77. doi: 10.1186/1471-2407-7-77. PMID 17488518